CLINICAL TRIAL: NCT01009346
Title: A Phase 1 Study of RAD001 in Combination w/ Cetuximab and Cisplatin as First-line Therapy in Recurrent & Metastatic Squamous Cell Cancer of the Head & Neck
Brief Title: RAD001 in Combination With Cetuximab and Cisplatin in Recurrent and Metastatic SCCHN
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Toxicity
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0916; NA_00023951 (Other: JHM IRB)
Record Dates: First submitted 2009-10-21; First posted 2009-11-06 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Everolimus; Cetuximab; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001 (Experimental): Daily RAD001 in combination with weekly cetuximab and cisplatin/ carboplatin on Day 1, 8 of each 28 day cycle.
  Interventions: Drug: RAD001; Drug: Cetuximab; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: RAD001 — Dose Level -1 2.5mg/day
  Dose Level 1 5mg/day*
  Dose Level 2 10mg/day
  MTD RAD001
  Other Names: Everolimus
Drug: Cetuximab — 250mg/m2/week
  Other Names: Erbitux
Drug: Cisplatin — 40mg/m2 Day 1, 8 every 28 days
  Other Names: cisplatinum; CDDP; cis-diamminedichloroplatinum(II)
Drug: Carboplatin — Carboplatin will be administered on Day1 and Day 8 of each 28 day cycle to a target AUC of 3 over 30 minutes. Carboplatin will be dosed using the Calvert formula:
  Total dose (mg) = (target AUC) x (glomerular filtration rate + 25) Creatinine clearance will be used to estimate the GFR. The Cockgroft-Gault formula will be used to estimate the creatinine clearance.
  Other Names: cis-Diammine(1,1-cyclobutanedicarboxylato)platinum(II)

SUMMARY:
1.Phase I: To estimate the Maximum Tolerated Dose (MTD) of RAD001 in combination with cetuximab and cisplatin for treatment of metastatic squamous cell cancer of the head and neck (SCCHN).

Secondary Objectives

1.To assess the toxicity of RAD001 in combination with weekly cetuximab and cisplatin on days 1 and 8 of each 28 day cycle in patients with recurrent or metastatic SCCHN,

DETAILED DESCRIPTION:
This was a dose escalation study with RAD001 in combination with cetuximab and cisplatin in recurrent/metastatic SCCHN. Patients with ECOG performance status 0-2, with no prior systemic therapy for recurrent/metastatic SCCHN were enrolled. The dose levels for RAD001 were 2.5mg, 5mg or 10 mg administered oral daily, cetuximab 250mg/m2 weekly infusion, and cisplatin 40mg/m2 days 1 and 8. Each cycle was 28 days. Safety monitoring plan was outlined in the protocol and study calendar at specific time points. Response was evaluated with CT/MRI and PET scans every 2 cycles. DLT criteria and MTD was defined.

Dose escalation followed the conventional 3+3 design.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed diagnosis of squamous cell carcinoma of the head and neck, with recurrent or metastatic disease.
2. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan. See Section 11 for the evaluation of measurable disease.
3. Patients must have had no prior monoclonal antibodies or small molecule tyrosine-kinase inhibitors for the treatment of recurrent or metastatic SCCHN. In addition, no prior chemotherapy for the treatment of recurrent or metastatic SCCHN is allowed.
4. If the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation. Patients must be greater than or equal to 12 weeks from completion of prior curative intent therapy including surgery, radiation, or systemic anticancer therapy. If palliative radiation therapy is given for recurrent or metastatic disease, patients must be greater than or equal to four weeks from treatment.
5. No concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix. Patients with prior history of malignancies must be disease free for greater than or equal to two years.
6. Age >18 years.
7. Life expectancy of greater than 4.5 months.
8. ECOG performance status <2 (Karnofsky >60%; see Appendix A).
9. Patients must have normal organ and marrow function as defined below:

   * leukocytes >3,000/mcL
   * absolute neutrophil count >1,500/mcL
   * platelets >100,000/mcL
   * total bilirubin less than or equal to 1.5 X institutional upper limit of normal or within normal institutional limits. or
   * AST(SGOT)/ALT(SGPT) <3.0 X institutional upper limit of normal - creatinine within normal institutional limits OR
   * creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal 3.1.8
10. As the investigational agent RAD001 requires enteral administration, patients must be able to receive adequate enteral nutrition by mouth or through a G-tube device.
11. The effects of RAD001 on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
12. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
2. Patients may not be receiving any other investigational agents.
3. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to RAD001 or other agents used in the study.
5. Patients receiving any medications or substances that are inhibitors or inducers of the isoenzyme CYP3A are ineligible. Lists including medications and substances known or with the potential to interact with the CYP3A isoenzymes are provided in the appendix.
6. Patients receiving chronic treatment with systemic steroids or other immunosuppressive agents are ineligible.
7. Patients with a known hypersensitivity to RAD001 (everolimus) or other rapamycin (sirolimus, temsirolimus) or its excipients.
8. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g. ulcerative disease; uncontrolled nausea, vomiting, or diarrhea; malabsorption syndrome or small bowel resection).
9. Patients with active bleeding diathesis or patients on oral anti-vitamin K agent (excluding low dose warfarin).
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, severely impaired lung function or psychiatric illness/social situations that would limit compliance with study requirements Severely impaired lung function is defined as spirometry and DLCO that is 50% of the normal predicted value and /or O2 saturation that is 88% or less on room air.
11. Pregnant women are excluded from this study because RAD001 is a mTOR inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with RAD001, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study.
12. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with RAD001. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shanthi Marur, MD, Principal Investigator — Johns Hopkins SKCCC
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Early Termination.
Pre-assignment Details: Early Termination
Period: Overall Study
Arm/Group | RAD001
Started | 9
Completed | 5
Not Completed | 4
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Groups:
- Study Arm: Drug: RAD001
  Other Names:
  Everolimus
  Dose Level -1 2.5mg/day
  Dose Level 1 5mg/day*
  Dose Level 2 10mg/day
  MTD RAD001 Drug: Cetuximab
  Other Names:
  Erbitux
  250mg/m2/week Drug: Cisplatin
  Other Names:
  cisplatinum CDDP cis-diamminedichloroplatinum(II)
  40mg/m2 Day 1, 8 every 28 days Drug: Carboplatin
  Other Names:
  cis-Diammine(1,1-cyclobutanedicarboxylato)platinum(II)
  Carboplatin will be administered on Day1 and Day 8 of each 28 day cycle to a target AUC of 3 over 30 minutes. Carboplatin will be dosed using the Calvert formula:
  Total dose (mg) = (target AUC) x (glomerular filtration rate + 25) Creatinine clearance will be used to estimate the GFR. The Cockgroft-Gault formula will be used to estimate the creatinine clearance.
Arm/Group | Study Arm
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.77778 (12.71591)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of RAD001 in Combination With Cetuximab and Cisplatin.
Description: MTD will be defined as a) the dose of RAD001 producing DLT in 0-1 out of 6 patients, or b) the dose level below the dose which produced DLT in <2 out of 6 patients, or c) the dose of 10mg po qd with less than 33% rate of DLT
Time Frame: 6 months
Population: Patients who received at least one cycle of RAD001 were included in the analysis.
Measure: Number; unit: mg
Groups:
- Study Arm (RAD001, Cetuximab, Cisplatin or Carboplatin): Phase I will be a single arm , dose finding study to determine the maximum tolerated dose (MTD) of daily RAD001 in combination with weekly cetuximab and cisplatin on Day 1, 8 of each 28 day cycle. The combination will be explored in successive cohorts of 3 patients each. The first cohort of 3 patients will receive doses corresponding to the first dose level. A full safety evaluation will be conducted when these patients have completed 8 weeks of therapy (2 cycles). If 0/3 patients treated at a dose level have a DLT, then a new cohort of 3 patients will receive treatment at the next dose level. If 1/3 patients have even one DLT, then 3 more patients will be treated at same dose level. If none of these patients has a DLT, then the next higher dose level will be administered to the next cohort of 3 patients; otherwise the inferior dose level will be considered the MTD. If >2/3 patients have a DLT, then the inferior dose level will be considered the MTD.
Arm/Group | Study Arm (RAD001, Cetuximab, Cisplatin or Carboplatin)
Number analyzed (Participants) | 7
mg | 10

2. Secondary Outcome: Progression Free Survival (PFS) of RAD001 in Combination With Weekly Cetuximab and Cisplatin.
Description: Median number of months for which participants are free of progression after initiating treatment with RAD001 in combination with weekly cetuximab and cisplatin.
Time Frame: 2 years
Population: Only 5 patients received at least one cycle of RAD001
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Study Arm (RAD001): Phase I will be a dose finding study to determine the maximum tolerated dose (MTD) of daily RAD001 in combination with weekly cetuximab and cisplatin on Day 1, 8 of each 28 day cycle. The combination will be explored in successive cohorts of 3 patients each. The first cohort of 3 patients will receive doses corresponding to the first dose level. A full safety evaluation will be conducted when these patients have completed 8 weeks of therapy (2 cycles). If 0/3 patients treated at a dose level have a DLT, then a new cohort of 3 patients will receive treatment at the next dose level. If 1/3 patients have even one DLT, then 3 more patients will be treated at same dose level. If none of these patients has a DLT, then the next higher dose level will be administered to the next cohort of 3 patients; otherwise the inferior dose level will be considered the MTD. If >2/3 patients have a DLT, then the inferior dose level will be considered the MTD.
Arm/Group | Study Arm (RAD001)
Number analyzed (Participants) | 5
months | 2.8 [1.6 to 13.9]

ADVERSE EVENTS:
Time Frame: 3 years.
Description: Early termination due to toxicity with the RAD001 in combination with cetuximab and cisplatin.
Groups:
- RAD001/Cetuximab/Cisplatin or Carboplatin: This was a dose escalation study with RAD001 in combination with cetuximab and cisplatin in recurrent/metastatic SCCHN. Patients with ECOG performance status 0-2, with no prior systemic therapy for recurrent/metastatic SCCHN were enrolled. The dose levels for RAD001 were 2.5mg, 5mg or 10 mg administered oral daily, cetuximab 250mg/m2 weekly infusion, and cisplatin 40mg/m2 days 1 and 8. Each cycle was 28 days. Safety monitoring plan was outlined in the protocol and study calendar at specific time points. Response was evaluated with CT/MRI and PET scans every 2 cycles. DLT criteria and MTD was defined.
Arm/Group | RAD001/Cetuximab/Cisplatin or Carboplatin
All-Cause Mortality (participants affected / at risk) | 9/9
Serious Adverse Events (participants affected / at risk) | 8/9
Other Adverse Events (participants affected / at risk) | 2/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001/Cetuximab/Cisplatin or Carboplatin (N=9)
GERD (Gastrointestinal disorders) | 1 (1)
Infusion Reaction (Cetuximab) (General disorders) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mucosal Edema (Laryngeal and Hypopharyngeal) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration (General disorders) | 1 (1)
Airway Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Septic Shock (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001/Cetuximab/Cisplatin or Carboplatin (N=9)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less